CLINICAL TRIAL: NCT06238986
Title: Relationship Between Alterations in the GI Microbiome and GI Inflammation on Symptom Burden in Women With Breast Cancer Receiving Chemotherapy
Status: Terminated | Type: Observational
Why Stopped: Lack of funding
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: MC230407; NCI-2024-00288 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 23-007468 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2024-01-25; First posted 2024-02-02 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Anatomic Stage I Breast Cancer AJCC v8; Anatomic Stage II Breast Cancer AJCC v8; Anatomic Stage III Breast Cancer AJCC v8

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational: Patients undergo stool and blood sample collection, complete questionnaires, and have their medical records reviewed on study.
  Interventions: Other: Non-Interventional Study

INTERVENTIONS:
Other: Non-Interventional Study — Non-interventional study

SUMMARY:
This study evaluates the relationship between alterations in the GI microbiome and GI inflammation on symptom burden in women with breast cancer receiving chemotherapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To describe changes in GI inflammation and the GI microbiome profile in women with breast cancer throughout chemotherapy.

II. To examine how GI inflammation and GI microbiome changes influence symptom experience is used above in women with breast cancer receiving chemotherapy.

III. To examine associations between microbial composition functional profiles at T1 and T2, T3 as well as T4 in patients who report symptom severity in neuropsychological and GI symptoms at the last three timepoints.

IV. To evaluate for differentially abundant metabolites and perturbed metabolic pathways associated with microbiome diversity in patients who do and do not report neuropsychological and GI symptom occurrence at T2, T3 and T4.

OUTLINE: This is an observational study.

Patients undergo stool and blood sample collection, complete questionnaires, and have their medical records reviewed on study.

ELIGIBILITY:
Inclusion Criteria:

* Female with a new diagnosis of breast cancer (stage I-III)
* Age 20 or older
* Able to read and write in English
* Chemotherapy naive and beginning the first cycle of moderately or highly emetogenic chemotherapy (For example, Taxotere + cyclophosphamide treatment +/- trastuzumab). Patients who have not received chemotherapy for five years or more are considered chemotherapy naive

Exclusion Criteria:

* Metastatic disease
* Cognitive impairment, based on clinician assessment, that would prevent completing measures
* Concurrent radiation therapy or radiation therapy within the last three months
* GI co-morbidities (i.e., irritable bowel syndrome, gastroesophageal reflux disease) or bowel surgery within the last three months
* A stoma preventing stool collection from the large intestine (i.e., ileostomy)

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with newly diagnosed stage I-III breast cancer recruited from the outpatient breast cancer clinic at University of Iowa Hospital and Clinics and at Mayo Clinic in Rochester and Mayo Clinic in Arizona.
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2024-03-22 (Actual); Primary Completion 2024-11-18 (Actual); Study Completion 2024-11-18 (Actual)

PRIMARY OUTCOMES:
Change in GI microbiome profile | Up to 1 month after chemotherapy treatment completion
  To examine longitudinal change in the GI microbiome, the coefficient of variation (CV) of alpha-diversity values will be calculated for stool samples. The CV represents the ratio of the standard deviation to the mean. A low CV indicates that an individual has relatively stable microbial diversity over time and a high CV indicates that an individual has higher microbial diversity over time.
Change in GI inflammation | Up to 1 month after chemotherapy treatment completion
  GI Inflammation will be quantified through measures of fecal calprotectin to indicate low, medium and high concentrations of bowel inflammation.
Symptom burden - MSAS | Up to 1 month after chemotherapy treatment completion
  Symptom burden will be measured with a modified version of the Memorial Symptom Assessment Scale (MSAS). The modified MSAS includes 41 symptom items, including 19 GI symptoms. Participants are asked to review the list of symptoms and indicate which had been present in the last week. For each symptom present, participants are asked to rate its duration, severity, and distress.
Symptom burden - MASCC-MAT | Up to 1 month after chemotherapy treatment completion
  Symptom burden will be measured with the Multinational Association of Supportive Care in Cancer-Antiemesis Tool (MASCC-MAT). The MASCC-MAT assesses acute (i.e., within 24 hours post-chemotherapy) and delayed (i.e., after 24 hours and up to 7 days post-chemotherapy) occurrence of chemotherapy-induced nausea (CIN).
Symptom burden - LFS | Up to 1 month after chemotherapy treatment completion
  Symptom burden will be measured with the Lee Fatigue Scale (LFS). The LFS consists of 18 items related to fatigue and energy. Scores range from 0-180 with higher scores indicating higher levels of fatigue.

SECONDARY OUTCOMES:
Associations between microbial composition functional profiles and symptom severity | Up to 1 month after chemotherapy treatment completion
  In patients who report symptom severity in neuropsychological and GI symptoms for at least three timepoints, stool samples will be tested to find distinct diversity and abundance changes between timepoints that are associated with symptom occurrence.
Change in metabolite abundance | Up to 1 month after chemotherapy treatment completion
  In patients who do and do not report neuropsychological and GI symptom occurrence for at least three timepoints, stool samples and blood samples will be evaluated using liquid chromatography-tandem mass spectrometry (LC-MS/MS) to evaluate for change in metabolite abundance and associations between bacterial composition and metabolic profiles.

CONTACTS AND LOCATIONS:
Overall Officials: Komal P. Singh, PhD, RN, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Rochester, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials